CLINICAL TRIAL: NCT04102462
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 764198 in Healthy Male Subjects (Double-blind, Randomised, Placebo-controlled, Parallel Group Design) and Effect of Food on the Relative Bioavailability of BI 764198 (Open-label, Randomised, Two-way Cross-over)
Brief Title: A Study to Test How Well Healthy Men Tolerate Different Doses of BI 764198
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1434-0007; 2019-002257-38 (EudraCT Number)
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Multiple rising dose part (Experimental)
  Interventions: Drug: BI 764198; Drug: Matching placebo
- Midazolam part (Experimental)
  Interventions: Drug: BI 764198; Drug: Matching placebo

INTERVENTIONS:
Drug: BI 764198 — Capsules
Drug: Matching placebo — Capsules

SUMMARY:
To investigate safety and tolerability of BI 764198 in healthy male subjects following oral administration of multiple rising doses per day over 14 days and to explore the pharmacokinetics (PK) of BI 764198 after single and multiple oral dosing. In addition, the effect of BI 764198 on the pharmacokinetics of midazolam, given as an oral microdose, will be explored after multiple oral dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects who meet any of the following criteria from administration of trial medication until 30 days after trial completion:

  * Males who are willing to use a medically acceptable method of contraception. Acceptable methods of contraception for use by male subjects include sexual abstinence, a vasectomy performed at least 1 year prior to dosing, and barrier contraception (condom)
  * Subjects who are not vasectomised or sexually abstinent have to ensure that an additional acceptable method of contraception will be used by his female partner such as intrauterine device (IUD), surgical sterilisation (including hysterectomy), hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to drug administration, or barrier method (e.g. diaphragm with spermicide)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days or 5 elimination half-lives, of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days or 5 elimination half-lives, of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more 24 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* A positive PCR test for SARS-CoV-2/COVID-19 or clinical symptoms suggestive for this disease at screening or within 2 days prior to admission to trial site (i.e. Day -3 to Day -2).
* further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug-related adverse events | Up to Day 34

SECONDARY OUTCOMES:
Multiple dose part - AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to Day 34
Multiple dose part - Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to Day 34
Multiple dose part - tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | Up to Day 34
Midazolam part - AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to Day 17
Midazolam part - Cmax (maximum measured concentration of the analyte in plasma) | Up to Day 17

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- [Derived] Schultz A, Halabi A, Seitz F, Lemmens K, Wulfrath HS, Lobmeyer MT, Retlich S, Choi W, Soleymanlou N. Phase 1 trials of BI 764198, a transient receptor potential channel 6 inhibitor, in healthy volunteers and participants with kidney impairment. Expert Opin Investig Drugs. 2025 May;34(5):415-423. doi: 10.1080/13543784.2025.2510673. Epub 2025 Jun 8. PMID 40455255